CLINICAL TRIAL: NCT06082011
Title: A Real-World Study to Evaluate the Clinical Performance and Safety of da Vinci SP Surgical System for Single-Port Gynecological Surgeries
Brief Title: A Real-World Study to Evaluate the Clinical Performance and Safety of da Vinci SP Surgical System for Single-Port Gynecological Surgeries(SPiM-RWS-GYN)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ISFMT-SP-004
Record Dates: First submitted 2023-09-19; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-08

CONDITIONS: Gynecological Surgeries
Keywords: radical hysterectomy; salpingectomy/oophorectomy; vaginal hysterectomy; total hysterectomy; myomectomy; ovarian cystectomy; deep endometriosis resection; pelvic and abdominal lymphadenectomy; sentinel lymph node resection by image development; uterus/vagino-sacral colpopexy; high uterosacral ligament suspension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- RWS study for SP Gynecological Surgeries: da Vinci SP Surgical System(SP1098)
  Interventions: Device: da Vinci SP Surgical System

INTERVENTIONS:
Device: da Vinci SP Surgical System — Model and specification: SP1098 Manufacturer: Intuitive Surgical, Inc.

SUMMARY:
Study name：A Real-World Study to Evaluate the Clinical Performance and Safety of da Vinci SP Surgical System for Single-Port Gynecological Surgeries Study purpose：This clinical trial is a real-world study to evaluate the clinical performance and safety of da Vinci SP Surgical System ("SP single-port robot" for short) for single-port robotic surgeries of gynecological benign and malignant tumors in the real world, providing a real world evidence for clinical application of the product in the Chinese population.

Study design：Retrospective + prospective, real-world study

English name: da Vinci SP Surgical System Model and specification: SP1098 Manufacturer: Intuitive Surgical, Inc.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients who have received or plan to receive gynecological surgeries with the SP single-port robot such as radical hysterectomy, salpingectomy/oophorectomy, vaginal hysterectomy, total hysterectomy, myomectomy, ovarian cystectomy, deep endometriosis resection, pelvic and abdominal lymphadenectomy, sentinel lymph node resection by image development, uterus/vagino-sacral colpopexy, and high uterosacral ligament suspension.
2. Patients who voluntarily participate in the study and sign the ICF (or exempt from signature of the ICF as approved by the EC).

Exclusion Criteria:

1. Patients with missing data on the primary endpoint in retrospective cases;
2. Patients having any contraindications of single-port robot surgery;
3. The intraoperative anatomy demonstrate that minimally invasive surgery is not suitable;
4. Patients who are considered inappropriate to participate in this Study by investigators.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have received or plan to receive single-port gynecological surgeries with the SP single-port robot such as radical hysterectomy, salpingectomy/oophorectomy, vaginal hysterectomy, total hysterectomy, myomectomy, ovarian cystectomy, deep endometriosis resection, pelvic and abdominal lymphadenectomy, sentinel lymph node resection by image development, uterus/vagino-sacral colpopexy, and high uterosacral ligament suspension.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint: Intraoperative conversion rate | Intraoperative
Primary safety endpoint: Incidence of device related or possibly related complications meeting the Clavien-Dindo Grading System level 3 or above criteria within 30 days after the surgery | 30 days

SECONDARY OUTCOMES:
Intraoperative bleeding volume | Intraoperative
Intraoperative blood transfusion rate | Intraoperative
Surgical duration | Intraoperative
Length of stay (LOS) | During the follow-up 1 day before discharge.The LOS is defined as the total inpatient days of each subject from the day of the surgery to the day of discharge (unit: days).
Admission to ICU and ICU LOS | During the follow-up 1 day before discharge, the admission to ICU and ICU LOS (unit: days) of each subject should be recorded.
Postoperative pain score | during the follow-ups 1 day (24±4 h), 3 days (72±4 h) and 1 month (30±5 days) after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai JiaoTong University School of Medicine affliated Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided